CLINICAL TRIAL: NCT06280287
Title: PET Imaging of Fibroblast Activation in Carotid and Coronary Atherosclerotic Disease
Brief Title: PET Imaging of Fibroblast Activation in Atherosclerosis
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FAPI-PLAQUE
Record Dates: First submitted 2024-01-17; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Carotid stenosis: Patients with carotid stenosis and suitable for carotid endarterectomy
  Interventions: Diagnostic Test: FAPI PET
- Coronary artery disease: Patients with stable ischemic heart disease or acute coronary syndrome
  Interventions: Diagnostic Test: FAPI PET

INTERVENTIONS:
Diagnostic Test: FAPI PET — 68Ga-FAPI PET/MR with high-resolution cardiovascular magnetic resonance vessel wall imaging for patients with carotid stenosis; 18FAl-FAPI PET/CT for patients with coronary artery disease

SUMMARY:
Fibroblast activation protein (FAP) is a fibroblast-specific marker expressed in atherosclerosis, associated with endothelial-to-mesenchymal transition and a rupture-prone plaque phenotype. This study aims to evaluate in-vivo fibroblast activation in carotid and coronary atherosclerotic diseases with FAPI PET and its correlation with histological vulnerability and clinical outcome.

DETAILED DESCRIPTION:
Fibroblast activation protein (FAP) is a fibroblast-specific marker expressed in atherosclerosis. Abundant FAP-expressing cells in atherosclerotic plaques co-express endothelial biomarkers involved in endothelial-to-mesenchymal transition. FAP upregulation is also associated with a rupture-prone plaque phenotype with a thin fibrous cap. Positron emission tomography (PET) with 68Ga-FAPI-04 has been demonstrated as a feasible method to image fibroblastic activation in the arterial wall. The current study aims to evaluate in-vivo fibroblast activation in carotid and coronary atherosclerotic diseases with FAPI PET and its correlation with histological vulnerability and clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* For the carotid stenosis group: patients with symptomatic carotid stenosis with >50% stenosis on carotid CTA; OR patients with unsymptomatic carotid stenosis with >70% stenosis on carotid CTA
* For CAD group: patients with stable ischemic heart disease OR acute coronary syndrome, including ST-elevation MId, non-ST elevation MI, and unstable angina
* signed informed consent

Exclusion Criteria:

* Pregnancy, lactation, or intention to become pregnant during the study
* Contradiction to MRI or CTA

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with carotid stenosis or CAD.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
SUVmax of atherosclerotic plaque in carotid or coronary arteries | through study completion, an average of 2 years
TBR of atherosclerotic plaque in carotid or coronary arteries | through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided